CLINICAL TRIAL: NCT01359904
Title: The Effect of Glucose Concentration in the Dialysate Bath on Glycemic Control Among Hemodialysis Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of Dialysis Glucose Bath on Glycemic Control in Hemodialysis (HD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Sameena Iqbal, Associate Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-361 GEN
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Results first posted 2016-11-28 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Type 2
Keywords: dialysate glucose; glycemic control; hypoglycemic episodes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Masking Description: no masking
Oversight: Data Monitoring Committee: No

ARMS (2):
- high dialysate bath (Active Comparator): additive is put in the dialysate to increase the concentration of glucose to 10mmol/l
  Interventions: Other: High Dialysate bath
- Standard dialysate glucose concentration (No Intervention): Standard 5.5 mmol/L dialysate glucose concentration.

INTERVENTIONS:
Other: High Dialysate bath — The dialysate bath assigned is 10mmol/L glucose, while the control group is assigned to 5.5 mmol/l glucose solution.
  Arms: high dialysate bath

SUMMARY:
Background:

Type II diabetes is a disease that affects more than 246 million people worldwide. Most importantly, one of the complications of type II diabetes is kidney damage and this has lead to many patients seeking hemodialysis treatment, a type of kidney replacement therapy. However, during hemodialysis treatment, many patients are greatly at risk for having their blood sugar drop below normal and this can lead to neurological problems. Also, it has been reported that hemodialysis patients who have poorer control of blood glucose levels are at risk to developing heart problems. It has been shown that adding 5.5 mmol/L of glucose in the hemodialysis treatment can reduce the chances of having an abnormal decrease in blood glucose levels. Currently, some institutions use 10 mmol/L of glucose (instead of 5.5 mmol/L) in the hemodialysis treatment, however, there is little documented support to justify for this action.

Objective:

The investigators are would like to explore the effects of use of 10 mmol/L of glucose in hemodialysis treatment and to determine if it worsens control of blood glucose levels, both during the treatment sessions and over the long term in type II diabetes patients. Also, patients on hemodialysis are prone to infection, so we will also observe if there is any change in infection rate among these patients with increased glucose in the treatment.

Methods:

The study will consist of 40 patients who will be randomly split into 2 groups. One group will be treated with 5.5 mmol/L glucose in the hemodialysis treatment and the other group will have 10 mmol/L glucose in the treatment. During the hemodialysis treatment, patient blood glucose will be measured at set intervals to check for any acute drops in glucose levels. Also, to assess long-term control of blood glucose levels, each patient will have 2 blood tests, one at the start and another at the end of the experiment. Signs of infection will be checked at the start of each session. Each patient will remain in their group for the duration of the study, which is 12 weeks.

DETAILED DESCRIPTION:
1. Study Design:

   Randomized-controlled study of all type 2 DM patients in dialysis to assess the effect of two different dialysate glucose concentrations, standard 5.5 mmol/L and high 10 mmol/L. The study period will be 20 weeks-4 weeks for recruitment, 12 weeks for the intervention and 4 weeks of data collection and analysis.
2. Study Population:

   All patients with diabetes type 2 in the Montreal General Hospital hemodialysis unit, will be identified by the Head nurses of dialysis units. The following patients will be excluded: anticipated to be transplanted within 6 months, expected death due to malignancy or severe infection within 6 months, uncontrolled blood sugars above 20mmol/l and unable to give consent due to neurologic reasons.

   Once the head nurse identifies the subject, the potential subject will be approached by the research assistant with a consent form.

   All patients will be consented by the research assistant through a written consent form. Then the subject will be randomly assigned to the standard or high glucose dialysate groups.
3. Methods

(i) Baseline Data collection for the standard or high glucose dialysate groups

The following demographic data will be noted: age, gender, duration of diabetes, duration of dialysis, comorbidity using Charlson Comorbidity index, vascular access type (arteriovenous fistula or permanent catheter) and cause of renal failure. The routine previous months' hemodialysis laboratory tests will be recorded such as complete blood count, serum electrolytes, serum glucose, calcium ionized or total, phosphate, parathyroid hormone levels, iron saturation, C reactive protein, ferritin, lipids and serum albumin. No additional blood tests will be taken. HbA1c values are taken every three months, therefore the intervention will be introduced after the HbA1c values have been taken within the month for the subject. No additional blood tests will be taken.

Blood pressure stability during the dialysis treatment will also be recorded defined as the differences in the pre and post mean arterial blood pressure will be documented in the last three dialysis treatments and their mean will be taken for each subject.

(ii) Intervention

After randomization, the subjects randomized to the high glucose group will be flagged in the hemodialysis orders, which on all electronic under the Nephrocare program. Similarly the standard glucose solution will also be flagged in the orders for the subjects randomized to that group.

(iii) Data collection during the Study

Both study groups will have a routine glucometer blood sugar test during the last hour of dialysis. The number of intradialytic asymptomatic and symptomatic hypoglycemic episodes will be recorded for each subject. Outcomes at the end of the 12 weeks of intervention: All subjects will have the following recorded:

1. Routine monthly blood work and the Hemoglobin A1c values
2. Number of episodes of serum glucose less than or equal to 3 mmol/L using the glucometer during dialysis treatments
3. Blood pressure stability during dialysis (mmHg)
4. Number of infection events during the 12 weeks will defined according to the Public Health Agency of Canada as stated below:

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 2 diabetes mellitus
* on chronic hemodialysis (for more than 3 months)
* age > 18 years

Exclusion Criteria:

* anticipated to be transplanted within 6 months
* expected death due to malignancy or severe infection within 6 months
* uncontrolled blood sugars above 20mmol/l
* unable to give consent due to neurologic reasons

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sameena Iqbal, MD, Principal Investigator — Associate Professor
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment occurred at 2 sites of McGill University Health Centre. The recruitment period was from June 1, 2011 to July 30, 2012.
Pre-assignment Details: Once the treating physician identified the potential subject, the potential subject was approached by the research assistant with a consent form.
  All patients were consented by the research assistant through a written consent form. Then the subject was randomly assigned to the standard or higher glucose dialysate groups.
Period: Overall Study
Arm/Group | High Dialysate Bath | Standard Dialysate Glucose Concentration
Started | 15 | 19
Completed | 14 | 19
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: forty subjects were needed to detect a difference in the mean change in the HbA1c from baseline to at the end of the study of 1% in the two dialysate concentration groups with a two-tailed t-test and variance of 1%, the required sample size will be 20 for each group with a power of 88% and alpha set at 0.05.
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dialysate Bath | Standard Dialysate Glucose Concentration | Total
Number analyzed (Participants) | 15 | 19 | 34
Age, Continuous [Median (Full Range); unit: years] | 73 [45 to 88] | 65 [35 to 87] | 71 [35 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 8 | 11 | 19
Region of Enrollment [Number; unit: participants]
  Canada | 15 | 19 | 34

OUTCOME MEASURES:

1. Secondary Outcome: Episodes of Hypoglycemia
Description: record number of episodes during dialysis with serum glucose below 4 mmol/L by glucometer
Time Frame: 3 months
Population: We planned forty subjects to detect a difference in the mean change in the HbA1c from baseline to at the end of the study of 1% among the two dialysate concentration groups with a two-tailed t-test and variance of 1%, the required sample size will be 20 for each group with a power of 88% and alpha set at 0.05.
Measure: Number; unit: episodes
Arm/Group | High Dialysate Bath | Standard Dialysate Glucose Concentration
Number analyzed (Participants) | 14 | 19
episodes | 2 | 10
Statistical Analysis 1: Comparison: High Dialysate Bath vs Standard Dialysate Glucose Concentration; Test type: Superiority or Other; p = 0.027, Chi-squared

2. Primary Outcome: Hemoglobin A1c Levels
Description: post intervention hemoglobin A1c levels
Time Frame: 3 months
Population: as for outcome 1
Measure: Median (Full Range); unit: percent
Arm/Group | High Dialysate Bath | Standard Dialysate Glucose Concentration
Number analyzed (Participants) | 14 | 15
percent | 7.1 [4.4 to 8.6] | 7.1 [4.7 to 10.4]
Statistical Analysis 1: Comparison: High Dialysate Bath vs Standard Dialysate Glucose Concentration; post intervention hemoglobin A1c levels; Test type: Superiority or Other; p = 0.67, Kruskal-Wallis

3. Secondary Outcome: To Record the Effects of a Higher Dialysate Concentration of Glucose on Glycemic Control of Hemodialysis Patients With Type 2 Diabetes Mellitus by Measuring Serum Levels of Hemoglobin A1c.
Description: Hemoglobin A1c levels will be measured before the intervention and after to assess any difference in the value. The blood samples were taken prior to dialysis treatments mid-week for each subject at baseline and at the end of the study in both the control and intervention groups.
Time Frame: 3 months
Measure: Median (Full Range); unit: percent
Arm/Group | High Dialysate Bath | Standard Dialysate Glucose Concentration
Number analyzed (Participants) | 14 | 19
percent | 0.3 [-2.2 to 2.6] | -0.1 [-2.6 to 1.1]
Statistical Analysis 1: Comparison: High Dialysate Bath vs Standard Dialysate Glucose Concentration; Test type: Superiority or Other; p = 0.20, Kruskal-Wallis

4. Secondary Outcome: the Number of Infections Related to Vascular Access in Dialysis Among Those Who Receive a Higher Glucose Concentration in the Dialysate and Those Who Receive the Standard Concentration
Description: In the two groups, we will measure the number of episodes of vascular access related infections ie. catheter, AV fistula or AV graft associated infections in the study period. The episode was defined as a diagnosis in the chart written by the nurse or physician with a prescription of antibiotics.
Time Frame: 3 months
Measure: Number; unit: episodes
Arm/Group | High Dialysate Bath | Standard Dialysate Glucose Concentration
Number analyzed (Participants) | 14 | 19
episodes | 4 | 3
Statistical Analysis 1: Comparison: High Dialysate Bath vs Standard Dialysate Glucose Concentration; Test type: Superiority or Other; p = 0.32, Chi-squared

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | High Dialysate Bath | Standard Dialysate Glucose Concentration
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/19
Other Adverse Events (participants affected / at risk) | 0/14 | 0/19

LIMITATIONS AND CAVEATS:
The study was only short term.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No